CLINICAL TRIAL: NCT04386330
Title: Firefighters Accessing Care for Trauma: A Clinical Case Series Testing the Efficacy of Distance-Delivered Narrative Exposure Therapy in Reducing PTSD/I Symptoms
Brief Title: Firefighters Accessing Care for Trauma: A Clinical Case Series of Distance NET for PTSD/I Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University of New Brunswick (Other)
Responsible Party: Principal Investigator, Patrick J. McGrath, Principal Investigator, IWK Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22081
Record Dates: First submitted 2020-05-08; First posted 2020-05-13 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Post Traumatic Stress Disorder; Post Traumatic Stress Injury
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Narrative Exposure Therapy (Experimental): Firefighters will receive distance-delivered NET administered by a paraprofessional.
  Interventions: Behavioral: Distance-delivered NET

INTERVENTIONS:
Behavioral: Distance-delivered NET — One-on-one intervention delivered by a paraprofessional; 12 weekly videoconference sessions at 90 minutes.

SUMMARY:
Repeated exposure to trauma is an unavoidable part of the job for firefighters. Because of this, many Canadian firefighters screen positive for posttraumatic stress disorder/injury (PTSD/I). Unfortunately, like the general population, firefighters face many barriers to accessing mental health care. As a result, additional efforts are needed to increase timely access to effective PTSD/I services that are delivered in a way that reduces confidentiality and stigma risk.

This research study will test the preliminary efficacy and feasibility of distance-delivered Narrative Exposure Therapy (NET) delivered by a paraprofessional for firefighters with PTSD/I. NET is an evidence-based intervention approach developed specifically for PTSD/I resulting from repeated and continuous trauma. The intervention will be conducted via videoconference with a trained paraprofessional supervised by a clinical psychologist. The NET intervention will consist of 12 weekly 90-minute videoconference sessions.

Approximately 25 firefighters will be recruited to participate in the study. To test the efficacy of the intervention, participants will complete self-report questionnaires about PTSD/I and other mental health symptoms pre- and post-intervention as well as two- and six-months following intervention completion. Participants will also complete an open-ended interview at the end of the intervention to assess feasibility and participant satisfaction.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet the following criteria to be eligible to move on to Consent

1. Be at least 19 years of age
2. Be able to understand spoken and written English at a Grade 8 level
3. Be employed, or have been employed, by the fire service or be current or past fire service volunteers.
4. Fulfill the criteria of full or subclinical PTSD/I according to the PCL-5.
5. Have access to a computer with Internet.
6. Live in Atlantic Canada or Ontario.
7. Consent to be audio- (for consent and interview) and video-recorded (for intervention sessions).

Exclusion Criteria:

1. Having a psychotropic medication change in the past three weeks.
2. Are currently engaged in or have previously been engaged in exposure therapy for PTSD/I.
3. Meet criteria for current mania or psychosis.
4. Endorse suicidal ideation with plan or intent.
5. Experience high levels of dissociation (as assessed by a score of >18.5 on the Shutdown Dissociation Scale).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in PTSD/I symptoms | Baseline, Immediately Post- intervention, 2 month follow up, 6 month follow up
  PTSD/I symptoms are measured with the PTSD Checklist - 5 (PCL-5)
Change in depressive symptoms | Baseline,Immediately Post-intervention, 2 month follow up, 6 month follow up
  Depression symptoms will be measured using the Patient Health Questionnaire (PHQ-9)
Disability | Baseline, Immediately Post-intervention, 2 month follow up, 6 month follow up
  Disability will be measured with the Sheehan Disability Scale

SECONDARY OUTCOMES:
Anxiety Symptoms | Baseline, Immediately Post-intervention, 2 month follow up, 6 month follow up
  Anxiety symptoms will be measured using the Generalized Anxiety Disorder - 7 item (GAD-7)
Physical Health | Baseline, Immediately Post-intervention, 2 month follow up, 6 month follow up
  Physical health will be measured with the Patient Health Questionnaire Physical Symptoms (PHQ-15)
Health Service Use | Baseline, Immediately Post-intervention, 2 month follow up, 6 month follow up
  Health service use will be measured using a series of questions regarding participant's use of health services as well as frequency and intensity of service use
Recruitment Rates | Baseline
  Recruitment rates will be tracked by research staff throughout the study
Intervention Adherence | Immediately Post-Intervention
  Intervention adherence will be measured via attendance records of participants kept by their coach. These attendance records will be used to measure the average number of completed sessions and the percentage of participants who did not complete the intervention.
Coach Alliance | Immediately Post-Intervention
  Coach alliance will be measured using the Working Alliance Inventory - Short Form Revised (WAI-SR)
Intervention Perceptions and Satisfaction | Immediately Post-Intervention
  Intervention perceptions and satisfaction will be measured via open-ended questions administered through a post-intervention interview

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Brunswick, Fredericton, New Brunswick, Canada

REFERENCES:
- [Derived] Olthuis JV, Kaltenbach E, Giberson E, Saryeddine T, Asmundson GJG, Carleton RN, Cramm H, Crombach A, Devlin J, Mack J, Lingley-Pottie P, Rao S, Sullivan M, Wozney L, McGrath PJ. Paraprofessional delivery of online narrative exposure therapy for firefighters. J Trauma Stress. 2023 Aug;36(4):772-784. doi: 10.1002/jts.22941. Epub 2023 Jun 8. PMID 37291963